CLINICAL TRIAL: NCT00584623
Title: Simultaneous Fluoroscopic and Endoscopic Examination of the Oropharyngeal Phase of Deglutition
Status: Withdrawn | Type: Observational
Why Stopped: Did not find interested patients.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200715188
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Dysphagia
Keywords: dysphagia; videofluoroscopy; flexible endoscopic evaluation
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To correlate findings between two commonly-used types of swallowing studies: videofluoroscopy and flexible endoscopic evaluation of swallowing (FEES).

DETAILED DESCRIPTION:
The specific aim of this study is to correlate findings between two commonly-used types of swallowing studies: videofluoroscopy and flexible endoscopic evaluation of swallowing (FEES). Specifically, the timing of swallowing events will be correlated between teh two studies. In addition, the pharyngeal constriction ratio (a validated measure of pharyngeal strength on videofluoroscopy) will be compared with the pharyngeal squeeze maneuver (an assessment of pharyngeal strength on FEES), with the hypothesis that there will be a strong correlation between PCR and pharyngeal squeeze.

ELIGIBILITY:
Inclusion Criteria:

* complaints of dysphagia
* scheduled to undergo videofluoroscopy
* able to tolerate both videofluoroscopic evaluation of swallowing and FEES

Exclusion Criteria:

* age less than 18
* contraindications to videofluoroscopy (reaction to barium, possible pregnancy)
* contraindications to FEES (bilateral obstructing nasal pathology or nasopharyngeal stenosis)
* specific/vulnerable populations (children, mentally handicapped, pregnant women, fetuses, prisoners, cognitive impairment, life-threatening disease, social or economic disadvantage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult clinic population in the UCD Otolaryngology Clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Belafsky, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States